CLINICAL TRIAL: NCT00919464
Title: Natural History of Anterior Compartment Pressures of the Thigh Following Femur
Brief Title: Natural History of Anterior Compartment Pressures of the Thigh Following Femur Fracture
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Michael Whitler, BS, IRB Admin, CAMC Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 06-04-1803
Record Dates: First submitted 2009-06-09; First posted 2009-06-12 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Femur Fracture
Keywords: Compartment pressure; compartment syndrome; femur fracture
MeSH Terms: conditions — Femoral Fractures; Compartment Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Needle Insertion into Femur (Other): Data gathering with monitoring of pressures in the thigh via via needle in femur.
  Interventions: Device: Pressure monitoring device; Device: Compartmental fracture pressure monitoring; Device: This small project is designed to be a non-randomized, investigational prospective trial of compartment pressures in the thigh following femoral fracture

INTERVENTIONS:
Device: Pressure monitoring device — monitoring device inserted to measure thigh compartment pressures
Device: Compartmental fracture pressure monitoring
Device: This small project is designed to be a non-randomized, investigational prospective trial of compartment pressures in the thigh following femoral fracture

SUMMARY:
This study is to determine the natural history of compartment pressures in the anterior thigh secondary to a fracture of the femoral shaft.

DETAILED DESCRIPTION:
Compartment syndrome is a painful condition where increased tissue pressure in a restricted area compromises circulation and endangers the tissue within that area possibly leading to surgery, amputation, major loss of function and in rare cases, death. Compartment syndrome of the thigh can be particularly devastating because of the size of the muscle and large amount of blood flow to the area, however it is one of the more rare and therefore least understood of all compartment syndromes. The purpose of this study is to determine the natural history of pressures of the anterior compartment of the thigh following femur fracture, which could help elucidate the diagnostic and treatment algorithms for thigh compartment syndrome. This small project is designed to be a non-randomized, investigational prospective trail to be conducted at the General Division of Charleston Area Medical Center. The target population consists of males and non-pregnant females age 18 and over who have suffered a mid-shaft femur fracture.

ELIGIBILITY:
Inclusion Criteria:

* femur fracture
* age 18 and older

Exclusion Criteria:

* patients who are not candidates for surgical repair of femur fracture
* patients not expected to survive more than 1 week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Compartment pressures | Pre-operative to 50 hours post operation

CONTACTS AND LOCATIONS:
Overall Officials: John DeLuca, MD, Principal Investigator — WVU Department of Surgery